CLINICAL TRIAL: NCT05458076
Title: A Phase 1, Randomized, Double-blind, Single-and Multiple-dose Escalation, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of QLS1128 and in Combination With Ritonavir in Healthy Participants
Brief Title: A Study of QLS1128 and in Combination With Ritonavir in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLS1128-101
Record Dates: First submitted 2022-07-06; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QLS1128 A-Dose 1~5 (Experimental): single dose
  Interventions: Drug: QLS1128 A-Dose 1~5 and Ritonavir
- QLS1128 C-Dose 1~3 (Experimental): Twice daily for 7 days
  Interventions: Drug: QLS1128 C-Dose 1~3 and Ritonavir
- QLS1128 D-Dose 1 (Experimental): fasting，high fat meal
  Interventions: Drug: QLS1128 D-Dose 1 and Ritonavir

INTERVENTIONS:
Drug: QLS1128 A-Dose 1~5 and Ritonavir — Cohort 1:
  QLS1128 A-Dose 1 or Placebo
  Cohort 2:
  Period 1: QLS1128 A-Dose 2 or Placebo, on day 1. Period 2:QLS1128 A-Dose 2 or Placebo with high fat meal on day 5. Period 3:QLS1128 A-Dose 2 or Placebo plus Ritonavir on day 9
  Cohort 3:
  QLS1128 A-Dose 3 or Placebo
  Cohort 4:
  QLS1128 A-Dose 4 or Placebo
  Cohort 5:
  QLS1128 A-Dose 5 or Placebo
  Arms: QLS1128 A-Dose 1~5
Drug: QLS1128 C-Dose 1~3 and Ritonavir — Cohort 6:
  Period 1: QLS1128 C-Dose 1 or Placebo, twice daily for 7 days. Period 2:QLS1128 C-Dose 1 or Placebo plus Ritonavir , twice daily for 7 days
  Cohort 7:
  Period 1: QLS1128 C-Dose 2 or Placebo, twice daily for 7 days. Period 2:QLS1128 C-Dose 2 or Placebo plus Ritonavir , twice daily for 7 days
  Cohort 8:
  Period 1: QLS1128 C-Dose 3 or Placebo, twice daily for 7 days. Period 2:QLS1128 C-Dose 3 or Placebo plus Ritonavir , twice daily for 7 days
  Arms: QLS1128 C-Dose 1~3
Drug: QLS1128 D-Dose 1 and Ritonavir — Cohort 9:
  Group A:QLS1128 D-Dose 1 plus Ritonavir under fasting condition, on day 1. QLS1128 D-Dose 1 plus Ritonavir under fatty food condition, on day 5
  Group B: QLS1128 D-Dose 1 plus Ritonavir under fatty food condition , on day 1. QLS1128 D-Dose 1 plus Ritonavir under fasting condition, on day 5
  Arms: QLS1128 D-Dose 1

SUMMARY:
A study to evaluate safety, tolerability and pharmacokinetics of QLS1128 sustained-release tablets and in combination with ritonavir tablets in healthy participants

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between ages of 18-45 years.
* Male subjects' weight ≥ 50 kg, female subjects' weight ≥ 45 kg; body mass index ≥ 19 kg/m2 and ≤ 27 kg/m2.
* Female participants of child-bearing potential/ Male subjects had fertile female partners must agree to use effective contraception from screening until 30 days after last dose.

Exclusion Criteria:

* Participant who have a past history of COVID-19 infection or are currently showing symptoms of COVID-19 infection.
* Participant who have been treated with any SARS-COV-2 neutralizing antibody or participated in clinical trials related to SARS-COV-2 (e.g., SARS-COV-2 neutralizing antibody, oral drug clinical trials, etc.).
* Participant who tested positive for SARS-COV-2 nucleic acid during the screening period, or who were positive for COVID-19 antibody if not vaccinated against COVID-19.
* Participant who have a clear history of allergy to drugs, food or pollen, or are allergic to ritonavir tablets and QLS1128 sustained-release tablets.
* Any clinical serious disease of cardiovascular, endocrine, neurological, digestive, respiratory, hematological, metabolic, psychiatric or other systems determined by the investigator may interfere with the results of this clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-07-03 (Actual); Primary Completion 2022-09-06 (Estimated); Study Completion 2022-09-06 (Estimated)

PRIMARY OUTCOMES:
The Adverse events of QLS1128 | Day 1 to Day 28
  Adverse events, including type, incidence, grade (determined with reference to NCI-CTCAE V5.0)

SECONDARY OUTCOMES:
The PK parameters of QLS1128 | Day 1 to Day 3
  Estimate of steady state Cmax for single dose administration of QLS1128

OTHER OUTCOMES:
The PK parameters of QLS1128 | Day 1 to Day 3
  Estimate of steady state AUC0-t for single dose administration of QLS1128
The PK parameters of QLS1128 | Day 1 up to Day 7
  Estimate of steady state Cmax for multiple dose administration of QLS1128
The PK parameters of QLS1128 | Day 1 up to Day 7
  Estimate of steady state AUC0-t for multiple dose administration of QLS1128

CONTACTS AND LOCATIONS:
Overall Officials: yunfei ju, M.D., Study Director — Qilu Pharmaceutical Co., Ltd.
Locations (1):
- Qilu Pharmaceutical Co., Ltd., Jinan, Shandong, China